CLINICAL TRIAL: NCT06236958
Title: Clinical Study on the Effect of Early Enteral Nutrition Implemented by Placing Nasojejunal Tube During Ovarian Cancer Surgery on Patients' Postoperative Recovery and Prognosis
Brief Title: Effect of Early Enteral Nutrition on Postoperative Recovery of Ovarian Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luo Chengyan (Other)
Responsible Party: Sponsor-Investigator, Luo Chengyan, chief physician, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Other Study IDs: 2023-SR-499
Record Dates: First submitted 2023-11-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Advanced Epithelial Ovarian Cancer
Keywords: Enteral Nutrition, Nasojejunal tube

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transnasal jejunal tube enteral nutrition group: Naso-jejunal tube was placed to the distal 15cm of Traitz ligament during the operation; short peptide enteral nutrient solution was heated by enteral nutrition pump and infused slowly and continuously 24 hours after the operation; during the period of infusion, the gastrointestinal tolerance of the patients was evaluated dynamically, and attention was paid to the absence of abdominal pain, diarrhea, constipation, vomiting, regurgitation, and misaspiration. According to the results of regular review of nutritional indicators, including hemoglobin, albumin, electrolytes, liver and kidney function, etc., increase the dosage of enteral nutrients in patients in appropriate amounts; patients with no abdominal distension after exhaustion and fluid intake, that is, the removal of nasojejunal tube, and replaced by oral intake of food.
  Interventions: Device: Transnasal jejunal tube
- Transvenous parenteral nutrition group: Nutrient solution was evenly titrated starting 24 hours after surgery. Configuration of nutritional solution: glucose and medium/long-chain fat emulsion as the main energy substances to provide calories, diabetic patients depending on the blood glucose level to adjust the pancreatic glucose ratio, and then assisted by subcutaneous injection of insulin to control blood glucose, if necessary, pay attention to the total amount of rehydration fluids, electrolytes, vitamins and micronutrient supplementation. Nutritional solution was evenly mixed in the laminar flow clean table and infused through the intravenous route, and oral feeding was started after exhaustion.
  Interventions: Other: Transvenous access

INTERVENTIONS:
Device: Transnasal jejunal tube — A naso-jejunal tube was placed in the operation, which is placed 15 cm below Traitz's ligament. A short-peptide enteral nutrient solution was heated by an enteral nutrient pump and infused into the patients within 24 hours after the operation. Before and at the end of the infusion, physiological saline was given to flush the tube, and at the end of the infusion, the catheter was closed to prevent liquid reflux and blockage of the tube. The catheter should be clamped shut at the end of the infusion. During the infusion period, the patient's gastrointestinal tolerance was dynamically evaluated. According to the results of a regular review of nutritional indicators, including hemoglobin, albumin, electrolytes, liver and kidney function, etc., increase the amount of enteral nutrients; remove the nasojejunal tube when the patient has no abdominal distension after exhaustion and feeding; and change to feeding through the mouth.
  Groups: Transnasal jejunal tube enteral nutrition group
Other: Transvenous access — A uniform drip of nutritional solution was started 24 hours postoperatively. Configuration of nutritional solution: glucose and medium/long-chain fat emulsion as the main energy substances to provide calories, calculated at 30 ~ 35 kcal/(kg-d), glucose-fat ratio is 6:4, pancreatic glucose ratio for those without a history of diabetes mellitus is 1:6 ~ 8, and for diabetic patients depending on the level of glucose, pancreatic glucose ratio is 1:3 ~ 4, and then assisted with subcutaneous injections of insulin to control glucose, if necessary. Pay attention to the total amount of rehydration fluid, electrolytes, vitamins, and trace elements supplemented. Mix the nutrient solution evenly in the laminar flow clean table and infuse it through the route at 2500~3000 ml/d; the infusion time is 8~12 h/d. After exhaustion, start to eat through the mouth.
  Groups: Transvenous parenteral nutrition group

SUMMARY:
This is a single-center, unblinded, prospective observational study, and the objective is to compare the effects of enteral nutrition via nasojejunal tube and parenteral nutrition via vein on patients' early recovery and prognosis who undergo tumor cytoreduction for ovarian cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the most lethal disease among gynecological malignancies, and its treatment is a comprehensive one mainly based on surgery. The perioperative nutritional status of patients affects their postoperative recovery, subsequent adjuvant therapy, and their prognosis. Hence, nutritional support therapy should be initiated for such patients in the early postoperative period to prevent further malnutrition. Conventional postoperative nutritional support therapy is performed through parenteral nutrition via vein, while the application of enteral nutrition via the nasojejunal tube in the postoperative period of ovarian cancer has not been reported in the literature. Therefore, in this study, the investigators took advantage of the characteristics of long surgical incisions and the wide surgical scope of ovarian cancer to investigate the effects of placing a nasojejunal tube during the operation and early enteral nutrition on postoperative recovery and prognosis in patients with advanced ovarian cancer, with the aim of accelerating the postoperative recovery of the patients, decreasing the incidence of postoperative complications, supplementing adjuvant chemotherapy in time, improving the survival outcome of the patients with advanced ovarian cancer, and providing gynecologists with a basis for enteral nutritional support therapy via nasojejunal tube after ovarian cancer surgery. In this study, the patients placed with a nasojejunal tube during the operation and enteral nutrition after the operation were included in the observation group, and the patients without a nasojejunal tube and parenteral nutrition after the operation were included in the control group. And the two groups were compared in terms of the indicators of postoperative recovery, the incidence of complications within the 30 days after operation, the cost of hospitalization, hospital stay, the interval between the operation and the first chemotherapy, the survival outcome, etc. The data involved in the study came from patient files, hospital databases, and long-term follow-up results.

ELIGIBILITY:
Inclusion Criteria:

* (1) The age is more than 18 years old and not more than 75 years old; (2) Ovarian cancer patients who are clearly diagnosed as epithelial ovarian cancer by pathological examination, whose tumors involve organs other than the pelvis as determined by preoperative imaging and intraoperative visual judgment, and who are at FIGO stage III or IV, and who undergo tumor cytoreductive surgery; (3) Patients without contraindication to nasoenteric tube placement and enteral nutrition; (4) Patients and their families were informed of the significance of the early use of enteral nutrition, precautions, adverse reactions, etc., before the operation, and they gave informed consent to this study and signed the informed consent; (5) Patients who received treatment in our hospital with complete clinical data.

Exclusion Criteria:

* (1) Patients with intestinal obstruction, severe intestinal infection, severe diarrhea, and acute abdomen right before surgery; (2) Patients with esophagogastric fundal varices and active gastrointestinal bleeding right before surgery; (3) Patients who undergo surgery to simultaneously resect the intestinal canal in the area more than 15cm distal to the ligament of Traitz; (4) Patients with severe cardiac, hepatic, and renal failure; (5) Patients with severe rhinitis, nasal mucous membrane damage, bleeding; (6) Patients with other malignant tumors combined within 3 months before surgery; (7) Metastatic ovarian cancer; (8) Those with missing clinical information; (9) Those with known hypersensitivity to enteral nutrition preparations.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the Department of Gynecology of the First Affiliated Hospital of Nanjing Medical University, aged 18-75 years old, with a definitive diagnosis of epithelial ovarian cancer by pathology, preoperative imaging, and intraoperative visual judgment of tumor involvement in organs other than the pelvic cavity, and FIGO Stage III or above, and proposed to undergo cytoreductive treatment of ovarian tumors.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | postoperative days 7, and 14
  To record the patient's hemoglobin on postoperative days 7 and 14 according to routine blood results
Intervals from surgery to the initiation of postoperative exhaustion and defecation | one month after surgery
  To record intervals from surgery to the initiation of postoperative exhaustion and defecation according to the medical record
The hospital stay after surgery and intervals from surgery to initiation of postoperative chemotherapy | one month after surgery
  To record the hospital stay after surgery and intervals from surgery to initiation of postoperative chemotherapy according to the medical record
The cost of hospitalization of peri operation | one month after surgery
  To record the cost of a patient's hospitalization of peri operation according to the medical record
Incidence of complications postoperative complications | one month after surgery
  To record the incidence of complications patient's postoperative complications for 30 days according to medical records, including: fever, intestinal obstruction, intestinal fistula, thrombosis, pulmonary embolism, poor incision healing, etc.
Quality of life scores | postoperative days 3
  To assess patients' quality of life scores on postoperative day 3 according to functional assessment of cancer therapy-ovary cancer (FACT-O) vision 4.0, with a minimum value of 0 and a maximum value of 156. The higher scores are, the better quality of postoperative survival is.
Serum sodium and potassium | postoperative days 7, and 14
  To record the patient's serum sodium and potassium on postoperative days 7 and 14 according to biochemical results.
Abnormal liver function | postoperative days 7, and 14
  To record the number of patients with abnormal liver function within 30 days postoperatively according to biochemical results. Abnormal liver function was defined as serum alanine aminotransferase and/or aspartate aminotransferase higher than 2.5 times the upper limit of normal values.
Abnormal renal function | postoperative days 7, and 14
  To record the number of patients with abnormal renal function within 30 days postoperatively according to biochemical results. Abnormal renal function was defined as serum creatinine and/or urea higher than 2.5 times the upper limit of normal values.
Serum albumin | postoperative days 7, and 14
  To record the patient's serum albumin on postoperative days 7 and 14 according to biochemical results.

SECONDARY OUTCOMES:
Survival outcomes | three years after surgery
  Survival outcomes at 3 years postoperatively, including progression, recurrence, death, and survival
Incidence of complications related to nasojejunal tubes | one month after surgery
  To record the incidence of complications related to tube placement in patients in the nasojejunal group according to medical records

CONTACTS AND LOCATIONS:
Overall Officials: Luo Chengyan, Doctor, Principal Investigator — The First Affiliated Hospital of Nanjing Medical University (Jiangsu Province Hospital)
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University (Jiangsu Province Hospital), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No